CLINICAL TRIAL: NCT06235931
Title: Prospective, Single-arm, Single-center Clinical Study of Darcilil Combined With AI Combined With Pyrrotinib in the Treatment of Elderly Advanced Triple-positive Breast Cancer.
Brief Title: A Clinical Study of Darcilil Combined With AI Combined With Pyrrotinib in the Treatment of TPBC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LK2023106
Record Dates: First submitted 2024-01-18; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Breast Neoplasms
Keywords: Triple-positive breast cancer; Dalsillie; Pyrrolizinib
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): Dalcilib +AI (letrozole/anastrozole/exemestane) + pyrrolizinib
  Interventions: Drug: Darcilide +AI (letrozole/anastrozole/Exemestane) + pyrrotinib

INTERVENTIONS:
Drug: Darcilide +AI (letrozole/anastrozole/Exemestane) + pyrrotinib — Darcilie: 125mg orally once a day, taken for 21 days and stopped for 7 days, 28 days as a cycle.
  AI: Letrozole: 2.5mg orally once daily, or anastrozole 1mg orally once daily, or exemestane 25mg orally once daily.
  Pyrrotinib: Initial dose of 240mg in the first week, if diarrhea and other side effects can be tolerated, 320 mg can be added in the second week, once a day, oral administration within 30 minutes after breakfast, 21 days for 1 cycle
  All investigational drugs should be used for disease progression or when patients have an intolerable adverse reaction or are withdrawn from the study for other reasons.
  Oral pyrrotinib is recommended along with prophylactic antidiarrheal medication. Antidiarrheal regimen 1: Oral imodium (2 tablets/times, 2 times a day) from the first week, 1 tablet, 2 times a day from the second week. Antidiarrheal regimen 2: montmorillonite powder (3 times a day, 1 pack/time)+ whole intestine sheng (3 pills/time 2 times a day).

SUMMARY:
Elderly patients with advanced triple-positive breast cancer have the characteristics of low physical status and poor treatment tolerance. Therefore, such patients are often unable to tolerate more toxic chemotherapy regimen, and it is particularly important to choose a highly effective and low-toxic treatment regimen. However, few studies have paid attention to the treatment of such patients in the past.

Pyrrotinib is a small molecule, irreversible, panerbb receptor tyrosine kinase inhibitor, which was independently developed by our country and has shown excellent efficacy in second-line anti-HER2 treatment of breast cancer, and has become the second-line standard treatment choice for advanced HER2-positive breast cancer. In addition, PHILA study results showed that the mPFS of pyrrotinib group reached 24 months. Compared with the control group, the duration of 10 months was significantly extended, indicating the significant efficacy of pyrrotinib in the first-line treatment of advanced HER2-positive breast cancer.

Darsili is a CDK4/6 inhibitor independently developed in China, which has been reconstructed and optimized in molecular structure, and has become a new CDK4/6 inhibitor with more powerful modification by introducing piperidine structure through replacement of classical electronic and other panbody. The results of DAWNA-2 study indicated that the mPFS of Dalsily combined AI group reached 30.6 months, which was significantly longer than 18.2 months of the control group, and was the longest in similar studies.

MUKDEN01 study, for the first time, tried the efficacy of pyrrotinib + letrozole + Dalsily regimen in the new adjuvant therapy of TPBC patients, and the results showed that ORR reached 87.4%, CR rate was 30.4%, and pCR rate was 35.4%. Therefore, to further confirm the efficacy and safety of this protocol in elderly patients with advanced triple positive breast cancer, we intend to conduct this study. This is a prospective, single-arm, single-center clinical trial in which participants were treated with darcilide +AI (letrozole/anastrozole/exemestane) + pyrrotinib until disease progression, toxicity became intolerable, informed consent was withdrawn, or investigator judgment required discontinuation. The successful development of this study provides a new direction for the first-line treatment of elderly advanced triple-positive breast cancer.

DETAILED DESCRIPTION:
In this open design, single-arm, single-center, prospective clinical study, 28 elderly patients with triple-positive advanced breast cancer were planned to receive treatment with darcilil combined with pyrrotinib and AI until the disease progressed, toxicity became intolerable, informed consent was withdrawn, or the investigator judged that the drug must be discontinued. The main objective of this study was to observe the safety and efficacy of Dalcilil combined with pyrrotinib and AI in the treatment of triple-positive senile advanced breast cancer.

In this study, the screening period did not exceed 28 days, and qualified subjects entered the study treatment period (every 28 days is a treatment cycle) after completing the screening examination and evaluation, and conducted the study treatment and visit according to the protocol. Imaging evaluation was performed according to the clinical routine during the study treatment. The imaging evaluation could be carried out according to the RECIST 1.1 standard, and the evaluation result of the investigator was the final result. At the end of treatment/withdrawal from the study, subjects should visit the research center to complete the corresponding safety check and imaging evaluation; In addition, a visit to the research center was conducted 28 days after the last treatment to complete the corresponding safety assessment.

Safety follow-up: the subjects were followed up until the initiation of other antineoplastic drugs. All AE recovered to grade 0-1 or baseline levels or died, whichever was achieved first.

Efficacy follow-up: All subjects were required to be followed until tumor progression or death or withdrawal of informed consent, whichever came first.

Follow-up for survival: All subjects were followed for survival until death or withdrawal of informed consent or the end of the trial, whichever came first.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age: ≥65 years old; 2. Histologically confirmed stage IV TPBC; 3. Without prior treatment, adjuvant endocrine therapy and anti-HER2 therapy should be completed for more than one year; 4.TPBC is defined as HER2-positive (3+ by immunohistochemistry, or 2+ by fluorescence in situ hybridization), ER-positive (more than 10% of tumor cells expressed estrogen receptor by immunohistochemistry), and PR-positive (at least 1% of tumor cells expressed progesterone receptor by immunohistochemistry) breast cancer; 5.ECOG score is 0-3 points; 6. Expected survival ≥12 weeks; 7. Normal function of major organs:

  1. Blood routine:

     Neutrophil (ANC) ≥1.5×109/L; Platelet count (PLT) ≥75×109/L; Hemoglobin (Hb) ≥90 g/L;
  2. Blood biochemistry:

     Total bilirubin (TBIL) ≤1.5× upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0×ULN; Alkaline phosphatase ≤2.5×ULN; Urea or urea nitrogen (BUN) and creatinine (Cr) ≤1.5×ULN;
  3. Heart color ultrasound:

Left ventricular ejection fraction (LVEF) ≥50%.

Exclusion Criteria:

* 1. Breast cancer with no evaluable lesions such as inflammation or occult; 2. Other malignancies within five years 3. Received other tyrosine kinase inhibitors, anti-HER2 treatment and T-DM1 treatment less than one year ago; 4. Patients with intestinal obstruction or fasting, gastrointestinal history, with diarrhea as the main symptom; 5. Suffering from mental illness or psychotropic substance abuse, unable to cooperate; 6. Pregnant or lactating women; 7. Participants considered unsuitable for inclusion by the researchers.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 34 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 29 months
  Defined as the date from enrollment until the first recording of tumor progression (as measured by RECIST 1.1 criteria, regardless of continuation of treatment) or the date of death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival | 29 months
  From the date of signing the informed consent to the date of death from any cause. For subjects who were still alive at the last follow-up, the OS was deleted based on the last follow-up time. For subjects who were lost to follow-up, the OS was calculated as the last confirmed survival time before the lost follow-up. The OS for data deletion is defined as the time from group entry to deletion.
Objective Response Rate | 29 months
  Proportion of all participants receiving investigational therapy who rated the best overall response (BOR) as complete response to CR or partial response to PR according to RECIST 1.1 criteria.
Disease Control Rate | 29 months
  Optimal proportion of subjects with CR, PR, and SD in overall response.
Objective Duration Of Remission | 29 months
  Defined as the period from the date of first recorded tumor remission (as measured by RECIST 1.1) to the date of first recorded objective tumor progression (as measured by RECIST 1.1) or the date of death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang P, Zhang Q, Tong Z, Sun T, Li W, Ouyang Q, Hu X, Cheng Y, Yan M, Pan Y, Teng Y, Yan X, Wang Y, Xie W, Zeng X, Wang X, Hu C, Geng C, Zhang H, Li W, Wu X, Zhong J, Xu J, Shi Y, Wei W, Bayaxi N, Zhu X, Xu B. Dalpiciclib plus letrozole or anastrozole versus placebo plus letrozole or anastrozole as first-line treatment in patients with hormone receptor-positive, HER2-negative advanced breast cancer (DAWNA-2): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2023 Jun;24(6):646-657. doi: 10.1016/S1470-2045(23)00172-9. Epub 2023 May 11. PMID 37182538
- [Result] Marty M, Cognetti F, Maraninchi D, Snyder R, Mauriac L, Tubiana-Hulin M, Chan S, Grimes D, Anton A, Lluch A, Kennedy J, O'Byrne K, Conte P, Green M, Ward C, Mayne K, Extra JM. Randomized phase II trial of the efficacy and safety of trastuzumab combined with docetaxel in patients with human epidermal growth factor receptor 2-positive metastatic breast cancer administered as first-line treatment: the M77001 study group. J Clin Oncol. 2005 Jul 1;23(19):4265-74. doi: 10.1200/JCO.2005.04.173. Epub 2005 May 23. PMID 15911866
- [Result] Wu J, Jiang Z, Liu Z, Yang B, Yang H, Tang J, Wang K, Liu Y, Wang H, Fu P, Zhang S, Liu Q, Wang S, Huang J, Wang C, Wang S, Wang Y, Zhen L, Zhu X, Wu F, Lin X, Zou J. Neoadjuvant pyrotinib, trastuzumab, and docetaxel for HER2-positive breast cancer (PHEDRA): a double-blind, randomized phase 3 trial. BMC Med. 2022 Dec 27;20(1):498. doi: 10.1186/s12916-022-02708-3. PMID 36575513
- [Result] Kaufman B, Mackey JR, Clemens MR, Bapsy PP, Vaid A, Wardley A, Tjulandin S, Jahn M, Lehle M, Feyereislova A, Revil C, Jones A. Trastuzumab plus anastrozole versus anastrozole alone for the treatment of postmenopausal women with human epidermal growth factor receptor 2-positive, hormone receptor-positive metastatic breast cancer: results from the randomized phase III TAnDEM study. J Clin Oncol. 2009 Nov 20;27(33):5529-37. doi: 10.1200/JCO.2008.20.6847. Epub 2009 Sep 28. PMID 19786670
- [Result] Huober J, Fasching PA, Barsoum M, Petruzelka L, Wallwiener D, Thomssen C, Reimer T, Paepke S, Azim HA, Ragosch V, Kubista E, Baumgartner AK, Beckmann MW, May C, Nimmrich I, Harbeck N. Higher efficacy of letrozole in combination with trastuzumab compared to letrozole monotherapy as first-line treatment in patients with HER2-positive, hormone-receptor-positive metastatic breast cancer - results of the eLEcTRA trial. Breast. 2012 Feb;21(1):27-33. doi: 10.1016/j.breast.2011.07.006. Epub 2011 Sep 8. PMID 21862331
- [Result] Niu N, Qiu F, Xu Q, He G, Gu X, Guo W, Zhang D, Li Z, Zhao Y, Li Y, Li K, Zhang H, Zhang P, Huang Y, Zhang G, Han H, Cai Z, Li P, Xu H, Chen G, Xue J, Jiang X, Jahromi AH, Li J, Zhao Y, de Faria Castro Fleury E, Huo S, Li H, Jerusalem G, Tripodi D, Liu T, Zheng X, Liu C. A multicentre single arm phase 2 trial of neoadjuvant pyrotinib and letrozole plus dalpiciclib for triple-positive breast cancer. Nat Commun. 2022 Nov 17;13(1):7043. doi: 10.1038/s41467-022-34838-w. PMID 36396665
- [Result] Zhang J, Meng Y, Wang B, Wang L, Cao J, Tao Z, Li T, Yao W, Hu X. Dalpiciclib Combined With Pyrotinib and Letrozole in Women With HER2-Positive, Hormone Receptor-Positive Metastatic Breast Cancer (LORDSHIPS): A Phase Ib Study. Front Oncol. 2022 Mar 7;12:775081. doi: 10.3389/fonc.2022.775081. eCollection 2022. PMID 35321427
- [Result] Spring LM, Gupta A, Reynolds KL, Gadd MA, Ellisen LW, Isakoff SJ, Moy B, Bardia A. Neoadjuvant Endocrine Therapy for Estrogen Receptor-Positive Breast Cancer: A Systematic Review and Meta-analysis. JAMA Oncol. 2016 Nov 1;2(11):1477-1486. doi: 10.1001/jamaoncol.2016.1897. PMID 27367583